CLINICAL TRIAL: NCT04141670
Title: Safety and Tolerability of S 48168 (ARM 210) for the Treatment of RYR1-related Myopathies (RYR1-RM)
Brief Title: S 48168 (ARM 210) for the Treatment of RYR1-related Myopathies (RYR1-RM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: RyCarma Therapeutics, Inc. (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institute of Nursing Research (NINR) (NIH); Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 200005; 1ZIANS003129-08 (NIH); Bench-to-bedside award 551673 (Other Grant/Funding Number: Intramural NINR)
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Results first posted 2024-04-19 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-02

CONDITIONS: RYR-1 Myopathy
Keywords: RYR1; Myopathy
MeSH Terms: conditions — Muscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Low dose group (Experimental): Experimental: 120 mg S48168 (ARM210; 6 x 20 mg tablets) daily for 29 days
  Interventions: Drug: S48168
- High dose group (Experimental): Experimental: 200 mg S48168 (ARM210; 10 x 20 mg tablets) daily for 28 days (1 participant) or 29 days (3 participants)
  Interventions: Drug: S48168

INTERVENTIONS:
Drug: S48168 — A novel oral small molecule which is designed to repair leaky RYR1 channels
  Other Names: ARM 210

SUMMARY:
This study proposes to test S 48168 (ARM210) in a Phase 1 trial in RYR1-RM patients, specifically. The objectives of this study are to explore the safety and tolerability, pharmacokinetics (PK), pharmacodynamics (PD)/target engagement (TE) of S 48168 (ARM210), as well as effects on muscle/motor function, and fatigue in RYR1-RM patients. The study population will include adult patients (≥18 years of age) who have demonstrated leaky RyR1 channels that are responsive to S48168 (ARM210) ex vivo.

DETAILED DESCRIPTION:
RYR1- related myopathy comprises a group of rare neuromuscular diseases. Affected individuals generally present with delayed motor milestones, muscle weakness, impaired ambulation, and, in severe cases, scoliosis, ophthalmoplegia, and respiratory distress all due to skeletal muscle weakness.

Causative variants in RYR1, which encodes the major calcium (Ca2+) release channel in skeletal muscle, RyR1, exert different effects on the RyR1 channel. They generally disrupt the normal Ca2+ flow between the sarcoplasmic reticulum (SR) and muscle cell cytosol and commonly result in excessive Ca2+ leak into the cytosol. Persistent Ca2+ leaks reduce its availability in the SR that is necessary for excitation-contraction coupling leading to the muscle weakness characteristic of this disease.

This open-label study consists of ten participants, randomized to two dose groups. All participants will have a diagnosis of RYR1-RM. In addition they have a prior muscle biopsy demonstrating a leaky RYR1 channel which responds to S48168 (ARM210) ex vivo. The first group of three participants will receive a low dose of S 48168 (ARM210) daily for 28 days. The second group of seven participants will receive a higher dose for 28 days. The decision to escalate to the higher dose will be made by an independent Data and Safety Monitoring Board (DSMB) after review of safety, tolerability and PK of the low daily dose. Safety and tolerability will be the primary objective in this study. In addition, exploratory objectives will include PK, PD/TE as well as measures of muscle/motor function and fatigue.

ELIGIBILITY:
INCLUSION CRITERIA:

Patients must meet all the following conditions to be eligible for enrollment into the study:

1. Body mass index (BMI) ≥ 18.0 and ≤ 36.0 kg/m2 at screening.
2. Confirmed genetic diagnosis of RYR1-RM and supporting clinical phenotype.
3. Ambulatory. Able to walk ten meters (with or without assistance e.g. with a cane).
4. Prior muscle biopsy with demonstrated leaky RyR1 channel.
5. Must have a CYP2C8 extensive or intermediate metabolizer genotype.
6. Daily use of medicines and dietary supplements need to be approved by the PI and Sponsor, or a drug/supplement-dependent wash-out prior to inclusion.
7. For male subjects: is sterile or agrees to use an appropriate method of contraception, including a condom with spermicide, from study drug administration on the first day of dosing until 5 half-lives plus 90 days (approximately 94 days) after the last dose of study drug administration. No restrictions are required for a vasectomized male subject provided the subject is at least 1-year post-bilateral vasectomy procedure prior to study drug administration on first day of the first dose. A male subject whose vasectomy procedure was performed less than 1 year prior to study drug administration on the first day of dosing must follow the same restrictions as a non-vasectomized male. Appropriate documentation of surgical procedure should be provided.
8. For male subjects: agrees to not donate sperm from study drug administration on the first day of dosing until 5 half-lives plus 90 days (approximately 94 days) after the last dose of study drug.
9. For female subjects of childbearing potential: uses one of the following highly effective birth control methods:

   * Prescribed hormonal oral contraceptives, vaginal ring, or transdermal patch.
   * Intrauterine device (IUD).
   * Intrauterine hormone-releasing system (IUS).
   * Depot/implantable hormone (e.g., Depo-provera®, Implanon).
   * Bilateral tubal occlusion/ligation.
   * Sexual abstinence:
   * Refraining from heterosexual intercourse during the entire period of risk associated with the study requirements.
   * If the participant decides to become sexually active during the study, then one of the highly effective birth control methods must be used.
10. For female subjects of non childbearing potential; defined by at least 1 of the following criteria:

    * Postmenopausal defined as 12 months of spontaneous amenorrhea and follicle stimulating hormone (FSH) serum level > 40mIU/mL. Appropriated documentation of FSH levels is required.
    * Surgically sterile by hysterectomy and/or bilateral oophorectomy with appropriate documentation of surgical procedure.
    * Has a congenital condition resulting in no uterus.
11. Willingness and ability to comply with scheduled visits, drug administration plan, laboratory tests, study restrictions, and study procedures (muscle biopsies and PK sampling).
12. Able to provide written informed consent and understands the study procedures in the informed consent form (ICF).

EXCLUSION CRITERIA:

The presence of any of the following conditions will exclude a patient from study enrollment:

1. Patient is mentally or legally incapacitated at the time of the screening visit or during the conduct of the study.
2. History or presence of alcoholism or drug abuse within the past 2 years prior to the first dose of study drug.
3. History or presence of hypersensitivity or idiosyncratic reaction to the study drug, related compounds, or inactive ingredients.
4. Positive urine drug or alcohol results at screening.
5. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C virus (HCV).
6. Patients with baseline ALT levels three times above the upper limits of normal (ULN) or baseline AST levels five times the ULN (isolated elevations of total bilirubin <2 X ULN with direct bilirubin below the ULN will be included).
7. Patients with severe pulmonary dysfunction at screening (Forced Vital Capacity (FVC) < 50% predicted) or evidence of pulmonary exacerbation. Pulmonary exacerbations refer to an acute worsening of respiratory symptoms that result from a decline in lung function.
8. Patients with a history of a seizure.
9. Subject has a history of cancer (malignancy) Exceptions: (1) Subjects with adequately treated non-melanomatous carcinoma or carcinoma in situ of the cervix may participate in the trial (2) Subjects with other malignancies who have been successfully treated > 10 years prior to the screening where in the judgment of the investigator has revealed no evidence of recurrence from the time of treatment through the time of the screening except those identified at the beginning of the exclusion criterion or (3) Subjects who in the opinion of the investigator are highly unlikely to sustain a recurrence for the duration of the trial.
10. Patients with uncontrolled diabetes defined as HbA1c > 7% or diabetic neuropathy.
11. Estimated creatinine clearance <40 mL/minute at screening, which may be calculated using the Chronic Kidney Disease Epidemiology Collaborative method (CKD-EPI), due to reduced muscle mass often seen in RYR1-RM patients.
12. Patients with a clinically significant abnormality on their ECG other than hypertensive related, or heart failure (ejection fraction <30%) or other clinically significant structural heart disease on echocardiogram.
13. Patients with a history of myocardial infarction in the last five years, or evidence of congestive heart failure.
14. Pregnant and breastfeeding women.
15. Patients who have taken Aspirin, Ibuprofen, or Naproxen within the 3 days prior to the muscle biopsy procedure, and/or patients who have taken Plavix (clopidogrel) or Brilinta (ticagrelor) 5 days prior to the muscle biopsy.
16. Unable to refrain from or anticipates the use of:

    * Any non-approved medicines and/or dietary supplements beginning 14 days prior to the first dose of study drug and throughout the study. Thyroid hormone replacement medication may be permitted if subject has been on same stable dose for the last 3 months prior to the first dose of study drug. Medicines that would contraindicate the skeletal muscle needle biopsy procedure, and therefore would be considered non- approved, include but are not limited systemic anticoagulants or oral direct thrombin inhibitors.
    * Any drugs known to be significant inducers or inhibitors of CYP2C8 enzymes for 28 days prior to the first dose of study drug and throughout the study. Any substrates of breast cancer resistance protein (BCRP).
17. Is currently taking any drug which raises gastric pH, including proton pump inhibitors or H2 antagonists. Antacids may be used if taken at night.
18. Donation of blood or significant blood loss within 56 days prior to the first dose of study drug.
19. Plasma donation within 7 days prior to the first dose of study drug.
20. Participation in clinical trials for other therapeutic investigational drugs simultaneously or within the 4 weeks prior to the first dose of study drug.
21. Ongoing medical condition that is deemed by the Principal Investigator to interfere with the conduct or assessments of the study or safety of the subject.
22. Is an NIH employee who is a subordinate/relative/coworker of a study investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Payam Mohassel, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: six months after publication
Access Criteria: published results and associated data will be available to academic medical researchers and patient advocacy groups upon request from ARMGO Pharma, INC

REFERENCES:
- [Derived] Todd JJ, Lawal TA, Chrismer IC, Kokkinis A, Grunseich C, Jain MS, Waite MR, Biancavilla V, Pocock S, Brooks K, Mendoza CJ, Norato G, Cheung K, Riekhof W, Varma P, Colina-Prisco C, Emile-Backer M, Meilleur KG, Marks AR, Webb Y, Marcantonio EE, Foley AR, Bonnemann CG, Mohassel P. Rycal S48168 (ARM210) for RYR1-related myopathies: a phase one, open-label, dose-escalation trial. EClinicalMedicine. 2024 Jan 25;68:102433. doi: 10.1016/j.eclinm.2024.102433. eCollection 2024 Feb. PMID 38318125

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose Group: Experimental:120 mg S48168 (ARM210; 6 x 20 mg tablets) daily for 29 days
  S48168: A novel oral small molecule which is designed to repair leaky RYR1 channels
Period: Overall Study
Arm/Group | Low Dose Group | High Dose Group
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Group | High Dose Group | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 3 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Body mass index [Mean (Standard Deviation); unit: kg/m^2] — ≥ 18.0 and ≤ 36.0 kg/m2 at screening.
  kg/m^2 | 24 (5) | 31 (5) | 28 (6)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Adverse Events When Treated With S48168 (ARM210)
Description: Composite safety and tolerability profile of S48168 (ARM210) based on adverse event reporting
Time Frame: 42 days
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Group | High Dose Group
Number analyzed (Participants) | 3 | 4
Participants
  Participants with fatal adverse events (all cause mortality) | 0 | 0
  Participants with serious adverse events | 0 | 0
  Participants with non-serious adverse events | 3 | 3

ADVERSE EVENTS:
Time Frame: Approximately two months
Arm/Group | Low Dose Group | High Dose Group
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 3/3 | 3/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose Group (N=3) | High Dose Group (N=4)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Headache (Nervous system disorders) | 0 (0) | 2 (2)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Mechanical utricaria (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-06-05): https://cdn.clinicaltrials.gov/large-docs/70/NCT04141670/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-28): https://cdn.clinicaltrials.gov/large-docs/70/NCT04141670/SAP_001.pdf